CLINICAL TRIAL: NCT01638884
Title: Cerebral Substrates of Prospective Memory in Healthy Young Adults and Disruptions in Normal Aging and Alzheimer Disease: a Study in Anatomical, Functional and Diffusion Tensor MRI.
Brief Title: Prospective Memory Imaging
Acronym: IMPRO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010-A00031-38
Record Dates: First submitted 2012-07-10; First posted 2012-07-12 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Alzheimer Disease
Keywords: Prospective Memory; Healthy Aging; Alzheimer Disease; Brain Imaging
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Young Healthy Subjects (Experimental)
  Interventions: Behavioral: Memory assessment; Other: Structural MRI; Other: Functional MRI; Other: Virtual reality / Memory assessment
- Middle age Healthy Subjects (Experimental)
  Interventions: Behavioral: Memory assessment; Other: Structural MRI; Other: Functional MRI; Other: Virtual reality / Memory assessment
- Elderly Healthy Subjects (Experimental)
  Interventions: Behavioral: Memory assessment; Other: Structural MRI; Other: Functional MRI; Other: Virtual reality / Memory assessment
- Mild Cognitive Impairment patients (Experimental)
  Interventions: Behavioral: Memory assessment; Other: Structural MRI; Other: Functional MRI; Other: Virtual reality / Memory assessment
- Alzheimer Disease patients (Experimental)
  Interventions: Behavioral: Memory assessment; Other: Structural MRI; Other: Functional MRI; Other: Virtual reality / Memory assessment

INTERVENTIONS:
Behavioral: Memory assessment — Neuropsychological tests including clinical and original tests to compare differences between each populations
Other: Structural MRI — to compare differences between each populations
Other: Functional MRI — to compare differences between each populations
Other: Virtual reality / Memory assessment — to compare differences between each populations

SUMMARY:
The purpose of this study is to investigate prospective merory (memory of intentions) in healthy controls and in aMCI (amnestic Mild Cognitive Impairment) and AD (Alzheimer Disease) patients.

ELIGIBILITY:
Inclusion Criteria :

* Education level > 7 years
* Native language: French
* Beck < 7
* Medical, neurological, neuropsychological and neuroradiological depth in accordance with the criteria for inclusion and exclusion-specific population, that is to say:

  * Young Healthy Subjects: between 18 and 44 years old;
  * Middle age Healthy Subjects: between 45 and 69 years old; without memory complaints, normal performances compared to the age and the educational level for all tests of the diagnostic battery.
  * Elderly Healthy Subjects: over 70 years old, without memory complaints, normal performances compared to the age and the educational level for all tests of the diagnostic battery.
  * MCI patients: over 50 years old, presenting the current criteria for amnestic MCI including: i) memory complaint, ii) deficits of the episodic memory (lower performance of at least 1 SD from the norm for age and cultural level for one or more scores of episodic memory and iii) normal performances compared to the age and the educational level of all other cognitive functions as memory, including tests to assess cognitive abilities.
  * Alzheimer's patients: over 50 years old, presenting the standard criteria of NINCDS-ADRDA probable Alzheimer's disease, including abnormal global cognitive function and deficits in at least two cognitive domains identified by the diagnostic battery and a mild to moderate Alzheimer's disease (MMSE ≥ 18).

Exclusion Criteria :

* The sudden onset of cognitive impairments (as opposed to their slow and gradual installation in Alzheimer's disease)
* A chronic neurological, psychiatric, endocrine, hepatic or infectious complaint
* A history of major disease (a lung, heart, metabolic, hematologic, endocrine disease or a severe cancer);
* A medication that may interfere with memory or metabolic measures
* A alcohol or drugs abuse
* claustrophobia, metallic object in the body
* A predominantly left-hand (score below 50% in Edinburgh Inventory).
* Protected adults, and persons not affiliated with a social security system will not participate in this study.
* Pregnant or suckling women
* The inclusion of a participant in another biomedical research protocol (during the study or within 12 months before inclusion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2010-09; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Rate of volume change of whole brain and other structural MRI measures | 1 Month
Cerebral regions implicated in prospective memory observed by functional MRI | 1 Month
Episodic memory as measured by Cognitive Tests | 18 Months
Virtual reality evaluation of prospective memory | 1 Month
Group differences for each imaging and neuropsychological measurement | 1 Month

CONTACTS AND LOCATIONS:
Overall Officials: Vincent de La Sayette, MD, Principal Investigator — University Hospital, Caen
Locations (3):
- France (3):
  - GIP Cyceron, Caen, Calvados
  - MRSH - University of Caen, Caen, Calvados
  - University Hospital Côte de Nacre, Caen